CLINICAL TRIAL: NCT05993546
Title: Randomized Controlled Trial of Miniaturized Percutaneous Nephrolithotomy With Vacuum-Assisted Access Sheaths Versus Conventional Sheaths for Treatment of Nephrolithiasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 23-104
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- vacuum-assisted sheath (Active Comparator)
  Interventions: Device: vacuum assisted sheath
- passive suction via conventional sheath (Active Comparator)
  Interventions: Device: passive suction via conventional sheath

INTERVENTIONS:
Device: vacuum assisted sheath — allows for simultaneous suction with continuous irrigation throughout the case to enhance visibility and facilitate stone retrieval
  Arms: vacuum-assisted sheath
Device: passive suction via conventional sheath — conventional access sheath for stone retrieval using current technique via passive suction
  Arms: passive suction via conventional sheath

SUMMARY:
The purpose of this study is to compare two variations of the mini-PCNL procedure using either a vacuum-assisted sheath or standard sheath which are both used for the surgical treatment of kidney stones. Both procedure types are commonly used in the treatment of kidneys stones and they have been shown to be safe and effective in the treatment of stones similar in size and location to your own.

DETAILED DESCRIPTION:
In this study we aim to compare two variations of the miniaturized percutaneous nephrolithotomy (Mini-PCNL) procedure which are both used for the surgical treatment of kidney stones. This procedure involves accessing the kidney via a small temporary tract that is placed through the patient's back during surgery. Both procedure types are commonly used in the treatment of kidneys stones and they have been shown to be safe and effective in the treatment of stones similar in size and location to your own.

Two procedure types will be investigated:

1. Miniaturized percutaneous nephrolithotomy performed using a 16 Fr (6 mm diameter) vacuum-assisted tube with suction capability to assess the kidney and extract the stone.
2. Miniaturized percutaneous nephrolithotomy performed using a 16 Fr (6 mm diameter) standard tube to assess the kidney and extract the stone.

Approximately 90 people will take part in this study at Cleveland Clinic. The duration of the study will include the day of the surgery and following hospital stay until postoperative follow-up appointment with the surgeon approximately 4-6 weeks after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned prone mini-PCNL and a preoperative NCCT
* Primary stone size: 10-25 mm
* Pre-existing indwelling nephrostomy tube or ureteral stent permitted
* Age: ≥ 18 years old
* Gender: all
* Ethnicity: all
* Capable of giving informed consent
* Capable and willing to fulfill requirements of the study

Exclusion Criteria:

* Anticoagulated or history of coagulopathy
* Congenital renal anomalies
* Prior ipsilateral upper urinary tract reconstructive procedures
* Conversion to open procedure
* Multiple access tracts
* Inability to give informed consent or unable to meet requirements of the study for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Stone free rate | 6 weeks
  The primary outcome of SFR will be measured using conventional follow up of post-operative NCCT at 6 weeks. NCCT provides the most definitive assessment for post-operative stone burden and allows assessment of radiolucent stones when compared to ultrasound or abdominal x-ray
Aim 2: Intraoperative variables | 3-7 days
  Patients with positive cultures will be treated with appropriate pre-operative antibiotics between 3 to 7 days depending on symptoms. Antibiotics on day of surgery will be selected according to their last pre-operative urine culture which is our standard of care for patients undergoing PCNL
Aim 3: Post-operative Outcomes and Complications | 1 day
  Post-operative pain scores will be evaluated using a visual analogue scale (VAS) in the post-anesthesia care unit (PACU) and on postoperative day 1. The questionnaire may be filled out on a paper survey or an electronic REDCap survey sent via email. An electronic VAS has shown to be reliable and interchangeable with a paper VAS

CONTACTS AND LOCATIONS:
Overall Officials: Sriharan Sivalingam, Principal Investigator — Principal Investigator
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States